CLINICAL TRIAL: NCT03676517
Title: Evaluation of Efficacy, Quality of Life and Cost Effectiveness of Short-course Radiotherapy Followed by Capecitabine Plus Oxaliplatin chemotheRapy and TME for High-risk Rectal Cancer (ESCORT Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0612
Record Dates: First submitted 2018-08-30; First posted 2018-09-18 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Intervention Model Description: Enrolled patient receive 1-week short-course radiation (5 Gy x 5) plus 6-week XELOX (capecitabine 1,000mg/m2 and oxaliplatin 130mg/m2 every 3 weeks) chemotherapy before total mesorectal excision (TME). Short-term outcomes including complications, TME completeness, and tumor response will be investigated. EORTC-QLQ-C30 questionnaire scoring will be used to evaluate QoL during the treatment period and after surgery. Cost effectiveness will be assessed using cost-utility analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative short-course radiotherapy (Experimental): 1-week short-course radiation (5 Gy x 5) plus 6-week XELOX (capecitabine 1,000mg/m2 and oxaliplatin 130mg/m2 every 3 weeks) chemotherapy before total mesorectal excision (TME)
  Interventions: Radiation: preoperative short-course radiotherapy

INTERVENTIONS:
Radiation: preoperative short-course radiotherapy — 1-week short-course radiation (5 Gy x 5) plus 6-week XELOX (capecitabine 1,000mg/m2 and oxaliplatin 130mg/m2 every 3 weeks) chemotherapy before total mesorectal excision (TME)

SUMMARY:
Multimodality treatment including surgery and radiotherapy is the current standard of care in locally advanced rectal cancer. Most clinical trials comparing short course radiotherapy (SCRT) with long course chemoradiotherapy(LCRT) did not find significant differences in oncological outcomes and short-term outcomes even though some debates. Recently, Stockholm III trial comparing SCRT plus delayed surgery with SCRT plus immediate surgery and LCRT demonstrated no differences with respect to short-term outcomes such as complications, mortality, and acute toxicity. However, overall quality of life (QoL) after curative treatment for rectal cancer is still major concern in both SCRT and LCRT. Furthermore, daily hospital visits for 5 weeks may be the cause of the increase of total medical cost due to indirect medical expense in patients with LCRT, especially in rural area. SCRT plus chemotherapy followed by delayed surgery may have the possibility of reducing total hospital costs as well as increasing QoL by proving non-inferiority in terms of perioperative outcomes. The present prospective single-arm phase 2 trial was designed to validate the efficacy, quality of life and cost effectiveness of preoperative short-course radiotherapy plus XELOX chemotherapy followed by delayed surgery for high-risk rectal cancer patient based on magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk patients of rectal cancer on pretreatment MRI using the following risk stratification system Location of the lower part of the tumor is measured below less than 10 cm on the anal verge and lower part of the tumor is located below the lower limit of the peritoneal reflection.

   If there is more than one, classify as a high risk group Positive CRM threatening: 5mm ≦ Extramural depth Positive EMVI.

   cN2: Positive Lateral pelvic LN metastasis
2. Between 19 and 80 years of age;
3. Satisfactory performance status: ECOG≦2
4. American Society of Anesthesiologists (ASA) physical status classification system class I~III
5. Adequate hematologic function: white blood cell(WBC) counts≥4,000/mm3, neutrophils counts ≥ 1,500/mm3, platelet counts ≥ 100,000/µL, hemoglobin ≥ 9g/L;
6. Adequate renal function: creatinine ≤ 1.5×upper normal limit

Exclusion Criteria:

1. The evidence of relapse of distant metastasis
2. Receiving treatment of other anti-cancer drug or methods
3. Patients have low compliance and are not able to complete the entire trial
4. Presence of uncontrolled life-threatening diseases
5. cT4 with infiltration of anterior organ on pretreatment MRI
6. cT4 with infiltration of internal or external anal sphincter on pretreatment MRI

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | Two weeks after surgery
  According to pathological response criteria, a total regression is considered a complete response

SECONDARY OUTCOMES:
Incidence of acute toxicities during radiation and chemotherapy | Three months
  Incidence of acute toxicities during radiation and chemotherapy
Incidence of surgical complications | Four weeks after surgery
  Incidence of surgical complications
Quality of life | Baseline and QOL at 8 weeks after radiotherapy
  QOL assessed using EORTC QLQ-CR29 survey form. The EORTC QLQ-CR29 is a 29-item colon and rectum cancer site-specific supplemental module that aims to enhance the sensitivity and specificity for colorectal cancer quality of life measures. The original English version comprises 4 multi-item scales (body image, urinary frequency, blood and mucus in stool, and stool frequency) and 17 functional/symptomatic single-items(anxiety, weight, sexual interest, urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problem, impotence or dyspareunia), with higher scores indicating better functional or worse symptomatic status. Of these 21 scales or items, only body image, anxiety, weight, and sexual interest are functional domain scales/items, and all the remaining are symptomatic.
Cost effectiveness | Three months
  QALYs (quality adjusted life years) with treatment protocol

CONTACTS AND LOCATIONS:
Locations (1):
- The Division of Colon and Rectal Surgery, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Lee JM, Lee J, Kim T, Kim NK, Cho MS. Long-Term Outcomes of Long-Course Chemoradiotherapy vs. Short-Course Radiotherapy Followed by Consolidation Chemotherapy in Rectal Cancer. Yonsei Med J. 2025 Dec;66(12):891-896. doi: 10.3349/ymj.2025.0216. PMID 41287502